CLINICAL TRIAL: NCT07081672
Title: The Effect of Interscalene Brachial Plexus Block Combined With General Anesthesia on Burst Suppression Ratio in Patients Undergoing Shoulder Surgery
Brief Title: Impact of Interscalene Block Combined With General Anesthesia on Burst Suppression in Shoulder Surgery Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bezmialem Vakif University (Other)
Responsible Party: Principal Investigator, Tugba KOK, MD, Bezmialem Vakif University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Screening
Other Study IDs: Tugba07
Record Dates: First submitted 2025-07-02; First posted 2025-07-23 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2025-07

CONDITIONS: Burst Suppression; Electroencephalogram; Interscalene Brachial Plexus Block
Keywords: burst supression; electroencephalogram; interscalene brachial plexus block; general anesthesia
MeSH Terms: interventions — Anesthesia, General; Control Groups

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: The study was conducted in a double-blind design: both the patients and the professional responsible for EEG data analysis were blinded to group allocation.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients in Group B received an ultrasound-guided interscalene brachial plexus block (ISB) (Active Comparator): A total of 20 mL of 0.125% bupivacaine was administered around the C5-C6 nerve roots under real-time ultrasound visualization. Fifteen minutes after the block, both sensory and motor block assessments were performed to confirm effectiveness. Following confirmation of a successful block, a standardized general anesthesia protocol was initiated using 1-2 mg/kg propofol, 1 mcg/kg fentanyl, and 0.6 mg/kg rocuronium, followed by endotracheal intubation. Anesthesia was maintained with sevoflurane (1.0-1.3 MAC), and depth of anesthesia was continuously monitored using the SedLine® EEG monitor.
  Interventions: Procedure: Ultrasound-guided interscalene brachial plexus block (ISB)
- Patients in Group K did not receive any regional anesthesia prior to general anesthesia induction. (Active Comparator): After standard monitoring was established, including ECG, non-invasive blood pressure, SpO₂, and SedLine® EEG monitoring, a 5-minute baseline EEG recording (Phase 0) was obtained with the patient at rest, eyes closed, and in a noise-minimized environment. Subsequently, general anesthesia was induced using 1-2 mg/kg propofol, 1 mcg/kg fentanyl, and 0.6 mg/kg rocuronium, followed by endotracheal intubation. Anesthesia was maintained with sevoflurane at 1.0-1.3 MAC in a mixture of 50% oxygen and air. To ensure adequate intraoperative analgesia, a remifentanil infusion (0.05-0.2 μg/kg/min) was administered and titrated according to Surgical Pleth Index (SPI) values, aiming to maintain SPI between 20-50.
  Interventions: Procedure: General Anesthesia (control group)

INTERVENTIONS:
Procedure: Ultrasound-guided interscalene brachial plexus block (ISB) — The intervention consisted of an ultrasound-guided interscalene brachial plexus block (ISB) administered to patients in Group B prior to general anesthesia. The block was performed using a posterior in-plane approach with real-time ultrasound visualization. A total of 20 mL of 0.125% bupivacaine was injected around the C5-C6 nerve roots under sterile conditions by experienced anesthesiologists.
  Arms: Patients in Group B received an ultrasound-guided interscalene brachial plexus block (ISB)
Procedure: General Anesthesia (control group) — General anesthesia without regional block
  Arms: Patients in Group K did not receive any regional anesthesia prior to general anesthesia induction.

SUMMARY:
This prospective, randomized, double-blind clinical study aimed to investigate the effects of combining general anesthesia with an interscalene brachial plexus block (ISB) on burst suppression ratio (BSR) and electroencephalographic (EEG) activity in patients undergoing elective shoulder surgery. A total of 50 patients were allocated into two groups: those receiving general anesthesia with ISB (Group B) and those receiving general anesthesia alone (Group K). Intraoperative EEG recordings were obtained from frontal electrodes (Fp1, Fp2, F7, F8) using a SedLine® monitor. Power spectral analysis was conducted for delta, theta, alpha, and beta frequency bands, alongside assessment of Patient State Index (PSI) and BSR.

DETAILED DESCRIPTION:
This prospective, randomized, double-blind clinical trial was conducted to evaluate the neurophysiological effects of combining interscalene brachial plexus block (ISB) with general anesthesia in patients undergoing elective shoulder surgery. The primary objective was to investigate how ISB influences intraoperative burst suppression ratio (BSR) and EEG-derived brain activity, using quantitative parameters such as power spectral densities of frequency bands and Patient State Index (PSI).

A total of 50 ASA I-III patients scheduled for shoulder surgery were randomly assigned into two groups: Group B (general anesthesia + ISB) and Group K (general anesthesia only). Standardized general anesthesia was maintained with sevoflurane in both groups. EEG data were recorded continuously using a SedLine® monitor from frontal electrodes (Fp1, Fp2, F7, F8) during four perioperative phases. Spectral analysis was performed using Fast Fourier Transform (FFT) and Welch's method to quantify power in the delta (0.5-4 Hz), theta (4-8 Hz), alpha (8-12 Hz), and beta (13-30 Hz) bands. BSR was calculated based on the duration of EEG suppression epochs, while PSI and SEF (Spectral Edge Frequency) were recorded continuously.

ELIGIBILITY:
Inclusion Criteria:

* Patients classified as ASA Physical Status I-III
* Aged between 18 and 65 years
* Scheduled for elective shoulder surgery under general anesthesia, with or without interscalene brachial plexus block

Exclusion Criteria:

* Advanced renal failure
* Advanced hepatic failure
* Body mass index (BMI) > 40 kg/m²
* History of central nervous system disorders
* Diagnosed psychiatric illness
* History of substance abuse
* Known allergy to any of the drugs used in the study
* Refusal to participate or to provide informed consent

Termination Criteria:

* Severe hypotension (mean arterial pressure < 50 mmHg despite treatment)
* Severe bradycardia (heart rate < 40 bpm requiring intervention)
* Profound hypoxia (SpO₂ < 90% despite oxygen support)
* Drug-related allergic reactions

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2025-01-29 (Actual); Primary Completion 2025-07-15 (Actual); Study Completion 2025-07-20 (Actual)

PRIMARY OUTCOMES:
Burst Suppression Ratio (BSR) | peroperative
  Burst Suppression Ratio (BSR): The main quantitative indicator of deep cortical suppression, calculated as the percentage of time the EEG signal remained in a suppression state (defined as amplitude <±10 μV for ≥0.5 seconds) during surgery. BSR was recorded continuously and analyzed across four perioperative phases (Phase 0-3).
Power Spectral Density (PSD) Analysis | peroperative
  The average spectral power (μV²) of EEG signals was analyzed for four conventional frequency bands-delta (0.5-4 Hz), theta (4-8 Hz), alpha (8-12 Hz), and beta (13-30 Hz)-using FFT-based spectral analysis. These values were calculated from frontal electrodes (Fp1, Fp2, F7, F8), and comparisons were made between Group B (ISB group) and Group K (control group) at each phase.
Patient State Index (PSI) | peroperative
  The Patient State Index (PSI), a proprietary quantitative measure ranging from 0 to 100, is derived from multichannel electroencephalogram (EEG) signals using the SedLine® brain function monitoring system. Higher PSI values indicate lighter levels of anesthesia or increased cortical activity, whereas lower values correspond to deeper anesthetic states. In this study, PSI values were utilized to monitor the level of consciousness and cortical stability during the intraoperative period. Particular emphasis was placed on PSI trends observed during Phase 1 (following the administration of the interscalene block but prior to the induction of general anesthesia), in order to investigate any pre-anesthetic central nervous system effects attributable to the regional block.

SECONDARY OUTCOMES:
Mean Arterial Pressure (MAP) | peroperative
  Intraoperative mean arterial pressure (MAP) was continuously monitored and recorded at predefined intervals throughout the procedure. Particular attention was paid to measurements taken during anesthesia induction, surgical positioning in the beach chair position, and skin incision. These data were analyzed to evaluate hemodynamic stability and to investigate the potential sympatholytic effects of the interscalene brachial plexus block (ISB).
Anesthetic and Analgesic Drug Consumption | peroperative
  Total doses of intraoperative sevoflurane, remifentanil, and propofol were recorded for each patient. Volatile anesthetic consumption was quantified in minimum alveolar concentration-hours (MAC-h). The aim was to evaluate whether ISB reduced the requirement for hypnotic and opioid agents during surgery.
Postoperative Pain Scores | During PACU stay (up to 2 hours)
  Postoperative pain intensity was assessed using the Numerical Rating Scale (NRS), which ranges from 0 (no pain) to 10 (worst imaginable pain). Higher scores indicate greater pain severity. Pain scores were recorded during the post-anesthesia care unit (PACU) stay, specifically within the first two hours following surgery, to evaluate early postoperative analgesia.
Nursing Delirium Screening Scale (NUDESC) | During PACU stay (up to 2 hours)
  The Nursing Delirium Screening Scale (NU-DESC) is a validated, nurse-administered tool used to detect signs of postoperative delirium. It assesses five domains: disorientation, inappropriate behavior, inappropriate communication, illusions/hallucinations, and psychomotor retardation. Each domain is scored from 0 to 2, resulting in a total score ranging from 0 to 10. A total score of ≥2 indicates a high probability of delirium. In this study, NU-DESC scores were recorded during the early postoperative period to identify any acute cognitive changes.
Heart Rate (HR) | peroperative
  Heart rate (HR) was continuously monitored intraoperatively and recorded at specified time points, with focused analysis during key phases such as anesthesia induction, patient positioning (beach chair position), and surgical incision. Group comparisons were made to assess ISB-associated modulation of cardiac autonomic response.
Oxygen Saturation (SpO₂) | peroperative
  Peripheral oxygen saturation (SpO₂) was monitored continuously during surgery and recorded at predetermined intervals. Measurements during critical phases, including induction, positioning, and incision, were evaluated to ensure adequate oxygenation and assess any indirect effects of ISB on respiratory function.

CONTACTS AND LOCATIONS:
Overall Officials: Kazım Karaaslan, MD, Study Director — Bezmialem Vakif University
Locations (1):
- Bezmialem Vakif University, Istanbul, Fatih, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No